CLINICAL TRIAL: NCT03414255
Title: A Phase 3, Prospective, Double-Blinded, Randomized Controlled Trial Of The Micronized dHACM Injection As Compared To Saline Placebo Injection In The Treatment Of Achilles Tendonitis
Brief Title: Micronized dHACM Injectable for the Treatment of Achille Tendonitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIAT001
Record Dates: First submitted 2018-01-23; First posted 2018-01-29 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2020-05

CONDITIONS: Tendonitis;Achilles
Keywords: Chronic Achilles Tendonitis
MeSH Terms: interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Micronized DHACM (Experimental): 1mL injection of 40mg Micronized dehydrated human amnion/chorion membrane (DHACM)
  Interventions: Biological: Micronized DHACM
- Saline Injection (Placebo Comparator): Injection of 1mL 0.9% Sodium Chloride Injection, USP
  Interventions: Drug: Saline Injection

INTERVENTIONS:
Biological: Micronized DHACM — 1 mL injection of 40mg Micronized dehydrated human amnion/chorion membrane (DHACM).
  Other Names: dHACM
  Arms: Micronized DHACM
Drug: Saline Injection — Injection of 1mL 0.9% Sodium Chloride Injection, USP
  Other Names: 0.9% NaCL; Normal Saline; Sodium Chloride Injection, USP
  Arms: Saline Injection

SUMMARY:
Prospective, Double-Blinded, Randomized Controlled Trial of the Micronized dHACM Injection as Compared to Saline Placebo Injection in the Treatment of Achilles Tendonitis

DETAILED DESCRIPTION:
Approximately 158 subjects will be enrolled in this study. Each patient will receive 1 injection and be evaluated for efficacy and safety during a 12 month observation period. Randomization will be 1:1. The study is expected to be completed in 24 months, inclusive of enrollment and follow-up of all subjects.

ELIGIBILITY:
Inclusion Criteria

All subjects enrolled must meet all the following criteria:

1. Confirmed diagnosis of Achilles tendonitis for ≥ 1 month (30 days) and ≤ 18 months by the investigator
2. VAS Pain scale of ≥ 45 at randomization
3. Achilles Tendonitis with conservative treatment for ≥1 month (30 days) while under the direction of the healthcare provider, including any of the following modalities:

   * Rest, Ice, Compression, Elevation (RICE)
   * Stretching exercises
   * Nonsteroidal Anti-inflammatory Drugs (NSAIDs)
   * Orthotics
4. Diagnostic AP and lateral X-Ray within 6 months of enrollment showing view of calcaneus negative for calcaneal fracture or structural abnormalities
5. BMI ≤ 40 kg/m2
6. Age from 21 to 80 years
7. Ability to sign Informed Consent and Release of Medical Information Forms
8. Ability to receive and respond to text messages or emails on a daily basis.

Exclusion Criteria Any potential subjects meeting any of the following criteria will be excluded from enrollment and subsequent randomization.

1. Prior surgery to the affected site.
2. Subjects requiring bilateral Achilles tendonitis treatment at time of enrollment
3. Prior use of any lower limb injection therapy, including corticosteroids or PRP in either limb within the last 3 months
4. Has diabetes either Type I or Type II
5. Systemic disorders associated with enthesopathy (disorder of entheses, i.e. bone attachments) such as Gout, Reiter's syndrome, rheumatoid arthritis, etc.
6. The presence of diagnosed comorbidities that can be confused with or can exacerbate the condition- to be assessed by X-ray - including but not limited to:

   * Calcaneal stress fracture
   * Suspected partial thickness tear of the Achilles tendon, as assessed by the investigator
   * Calcaneal tumor
   * Tarsal tunnel syndrome (diagnosed)
   * Significant bone deformity of the foot that may interfere with the study
7. The presence of diagnosed comorbidities that require surgery or are unlikely to improve - to be assessed by Investigator-including but not limited to:

   * Nerve entrapment syndrome
   * Acute traumatic rupture of the Achilles tendon
   * Partial thickness tears of the Achilles Tendon
8. Affected site exhibits clinical signs and symptoms of infection
9. Known allergy or known sensitivity to Aminoglycosides
10. Subjects who are non-ambulatory
11. History of more than 14 days of treatment with immune-suppressants (including systemic corticosteroids) or cytotoxic chemotherapy within 30 days prior to enrollment, or who are anticipated to require such medications during the course of the study
12. Prior radiation at the site
13. Use of any investigational drug(s) or therapeutic device(s) within 3 months preceding enrollment
14. Immune system disorders including Systemic Lupus Erythematosus (SLE), Fibromyalgia, Acquired Immunodeficiency Syndrome (AIDS), Human Immunodeficiency Virus (HIV) or Lyme disease
15. History of any conditions (including drug or alcohol abuse, medical or psychiatric condition) that is likely to impair understanding of or compliance with the study protocol, in the judgment of the investigator
16. Pregnancy at enrollment or within last 6 months, women who are breastfeeding, or women of childbearing potential who are planning to become pregnant during the time of the study OR are unwilling/unable to use acceptable methods of contraception (birth control pills, barriers, or abstinence)
17. Workers' compensation patients

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Change in VAS score | 90 days
  Visual Analog Scale, Left end point is "No Pain". Right end point is "worst pain imaginable"
Incidence of adverse events | 365 days
  The incidence of related Adverse Events (AEs), Serious Adverse Events (SAEs), and Unanticipated Adverse Events during the first 12 months post injection

SECONDARY OUTCOMES:
Foot Function Index Revised (FFI-R) (Short Form) | 90 days
  Subjects circle the number that correlates how bad their foot pain was in certain situation.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Miller, MD, Principal Investigator — MedStar Union Memorial Hospital Baltimore, MD
Locations (14):
- United States (14):
  - Central Research Associates, Birmingham, Alabama
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - ILD Research Center, Carlsbad, California
  - Foot and Ankle Clinic, Los Angeles, California
  - Five Cities Foot Clinic, Pismo Beach, California
  - South Florida Veterans Affairs, Miami, Florida
  - Doctors Research Network, Miami, Florida
  - Northside Podiatry, Buford, Georgia
  - Foot and Ankle Center of Illinois, Springfield, Illinois
  - Advanced Foot & Ankle Center, Las Vegas, Nevada
  - University Orthopedics Center, Altoona, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Futuro Clinical Trials, McAllen, Texas
  - Coastal Podiatry, Inc., Virginia Beach, Virginia